CLINICAL TRIAL: NCT05953909
Title: Efficacy and Safety of Eribulin-Based Regimen in the Treatment of Metastatic Triple-Negative Breast Cancer and Comparison With Other Chemotherapy Regimen: A Single-Center Retrospective Study
Brief Title: A Study of Eribulin-Based Regimen Versus Other Chemotherpy in Triple-Negative Metastatic Breast Cancer (ERI-Based-01).
Acronym: ERI-Based-01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: K2023-079-01
Record Dates: First submitted 2023-05-17; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Eribulin-Based Regimen: Not Applicable since observational study
  Interventions: Drug: Eribulin-Based Regimen; Drug: nab-paclitaxel based regimen; Drug: Other Chemotherapy Regimen
- nab-paclitaxel based regimen: Not Applicable since observational study
  Interventions: Drug: Eribulin-Based Regimen; Drug: nab-paclitaxel based regimen; Drug: Other Chemotherapy Regimen
- Other Chemotherapy Regimen: Not Applicable since observational study
  Interventions: Drug: Eribulin-Based Regimen; Drug: nab-paclitaxel based regimen; Drug: Other Chemotherapy Regimen

INTERVENTIONS:
Drug: Eribulin-Based Regimen — Eribulin Mesylate will be administered as a 1.4 mg/m^2 intravenous (IV) injection over 2 to 5 minutes on day 1 and day 8 of each 21-day cycle until unacceptable toxic effects or disease progression or other termination criteria appeared. Patients received up to two years of treatment.
  Other Names: Not Applicable since observational study
Drug: nab-paclitaxel based regimen — nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and carboplatin given IV at AUC 5 on days 1 every 21 days x 6 cycles.
  Other Names: Not Applicable since observational study
Drug: Other Chemotherapy Regimen — TX：Docetaxel 75mg/ m^2 D1 Q3W (or paclitaxel 175mg/ m2 D1 Q3W)+Capecitabine 850-950mg/ m^2, BID D1-14, Q3W.
  GP:Gemcitabine 800-1000mg/ m^2, D1,8 Q3W+Cisplatin 75mg/m^2, D1-3, Q3W. AT:Epirubicin 75mg/ m 2, D1, Q3W+Docetaxel 75mg/ m^2 D1 Q3W (or paclitaxel 175mg/ m^2 D1 Q3W)
  T:Docetaxel 75mg/ m ², D1 Q3W (or paclitaxel 80mg/ m ² QW)
  Other Names: Not Applicable since observational study

SUMMARY:
A Single-Center Retrospective Study About Efficacy and Safety of Eribulin-Based Regimen in the Treatment of Metastatic Triple-Negative Breast Cancer and Comparison With Other Chemotherapy Regimen

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70.
2. The pathologic diagnosis of unresectable recurrent or metastatic triple-negative breast cancer ［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
4. Patients with at least one measuring lesion that was conformed to RECIST v1.1 standard.
5. Patients receiving eribulin-based therapy received at least two cycles of eribulin-based chemotherapy. Eribulin was treated until disease progression, unacceptable toxicity or patient refusal of treatment.
6. Adverse events were recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE 5.0).

Exclusion Criteria:

1. Patients previously treated with eribulin.
2. Patients with grade ≥3 adverse events did not recover according to CTCAE 5.0 criteria.
3. Not applicable to combined chemotherapy, or allergic or intolerant to related drugs.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pathologic diagnosis is unresectable recurrent or metastatic triple-negative Chinese Breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free surviva (PFS) | up to 24 months
  The interval from the date of randomization to the first imaging confirmed progression of disease or death from any cause.
Overall survival (OS) | up to 24 months
  The time interval from the date of randomization to death due to any cause.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients
Disease Control Rate (DCR) | 12 months
  According to recist1.1 standard, the proportion of patients whose best remission was CR, PR or SD accounted for the total number of evaluable patients.
Incidence of adverse events | 12 months
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: weiwei Huang, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China